CLINICAL TRIAL: NCT02442115
Title: The MET Signaling System, Autism and Gastrointestinal Dysfunction
Brief Title: Impact of Improving Gastrointestinal Symptoms on Autism Symptoms and Oxidative Stress
Status: Completed | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Pat Levitt, PhD, Simms/Mann Chair in Developmental Neurogenetics, Institute for the Developing Mind, Children's Hospital Los Angeles
Other Study IDs: CCI-09-00212
Record Dates: First submitted 2015-03-25; First posted 2015-05-13 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Autistic Disorder; Constipation; Gastrointestinal Diseases
Keywords: Autism; Autism Spectrum Disorder (ASD); Tummy Troubles; Constipation; GI Disorders; Gastrointestinal Disorders; Gastrointestinal; Oxidative Stress; Stomach problems; Behaviors; Autistic; ASD; MET gene; GID; Pediatric; Pediatric GI disorders; Children with Autism; functional constipation
MeSH Terms: conditions — Autistic Disorder; Constipation; Gastrointestinal Diseases; Autism Spectrum Disorder; Digestive System Diseases; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine sample collection. Saliva sample collection for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD with GID: Children with Autism Spectrum Disorder with Functional Constipation will be treated with standard of care defined by NASPGHAN by a pediatric gastroenterologist, and evaluated at 4 visits over 1 year for their medical condition. These children will be enrolled in some ASD treatment program by their parents. The treatment program is not part of the current study. Measures of ASD symptoms will be done at each visit to determine social communication, emotional and cognitive improvement due to the FC treatment. Measures of F2-isoprostane, a marker of oxidative stress, will be done at each visit to determine if FC treatment and ASD symptom improvement relates to improvement in a child's physiology.
  Interventions: Other: Treatment of Functional Constipation by
- ASD without GID: Children Autism Spectrum Disorder without Functional Constipation will be evaluated for their ASD symptoms at 4 times over 1 year. These children will be enrolled in some ASD treatment program by their parents. The treatment program is not part of the current study. Measures of F2-isoprostane, a marker of oxidative stress, will be done at each visit to determine if ASD symptom improvement relates to improvement in a child's physiology.

INTERVENTIONS:
Other: Treatment of Functional Constipation by — The NASPGHAN protocol is used by pediatric gastroenterologist to treat functional constipation. Status is monitored at 4 visits and adjustments to treatment are made based on clinical standards and judgment.
  Other Names: NASPGHAN standard of care
  Groups: ASD with GID

SUMMARY:
The clinical manifestation of autism spectrum disorder (ASD) is complex, with medical and mental health disruptions that occur with the three core behavioral criteria used for diagnosis (social behavior, communication, restricted interests/repetitive behavior). Co-occurring medical conditions, such as gastrointestinal dysfunction (GID), often are overlooked when designing research strategies to understand the mechanisms underlying the expression of ASD. This study was initially a collaboration between Children's Hospital Los Angeles (CHLA) and the Children's Hospital at Vanderbilt University. The current research project proposes to recruit subject at CHLA and the Center for Autism and Developmental Disorders (CAND), a Children's Hospital of Orange County and University of California Irvine (UCI) Health collaborative program. In Aim 1, the investigators will characterize GID in pediatric populations with ASD. Over a 12 month period, subjects will receive standard of care for their GID, typically functional constipation. The study population will be characterized with a standardized instrument for diagnosing functional GI disorders in children, the Questionnaire on Pediatric Gastrointestinal Symptoms, and with the clinical acumen of an experienced pediatric gastroenterologist. Nutritional information also will be collected to determine whether there are patterns of GIDs that correlate with dietary and nutritional status. The in-depth characterization and treatment of GIDs in children with ASD will provide a unique way of determining if ASD symptom and GID symptom improvement are related to each other. In Aim 2, the investigators will do in-depth assessment of each subjects functional status for social communication, emotional regulation, cognitive function, speech-language, sensory integration, and a biomarker of oxidative stress. The latter will be measured in urine samples over the course of one year. There are no direct interventions for autism symptoms in this study. Rather, subjects will receive standard of care for the GID diagnosis and secondary effects on ASD symptoms will be evaluated. Our power calculation shows that the investigators will be adequately powered with the proposed study design and recruitment targets. As part of the study, the investigators have developed a collaboration with investigators in the University of Southern California (USC) School of Engineering, in which the investigators will work with them to develop computational tools to assist in the characterization of videotaped Autism Diagnostic Observation Schedule (ADOS-2) assessments.

DETAILED DESCRIPTION:
Children ages 7 years 0 months to 12 years 11 months will be recruited into 1 clinical group (ASD+/FC+), utilizing the following clinics in Southern California:

CHLA-affiliated Clinics

* Boone-Fetter Clinic, home of the CHLA Autism Treatment Network
* University Center of Excellence on Developmental Disabilities (UCEDD) Clinic at CHLA - UC Irvine/Orange County-affiliated clinics
* Center for Autism and Neurodevelopmental Disorders in Orange County
* Children's Hospital of Orange County Exclusion criteria include a diagnosed syndromic disorder, prematurity, failure to meet standard birth weight, not enrolled in any ASD treatment program. For each child, the Questionnaire on Pediatric Gastrointestinal Symptoms (QPGS)-Rome III is administered and the child is seen by a board-certified pediatric gastroenterologist. The child will be seen at baseline, 3, 6 and 12 months for their research visits. Treatment of FC in children with ASD is based on the Autism Treatment Network (ATN) modified protocol of the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN) and includes the following: 1) a thorough dietary history is reviewed and adjusted for introducing a diet rich in fiber (or supplements if able to be tolerated by the child; typically this will be in older children in the study); 2) assessment of abdominal pain, perianal skin tags, hemorrhoids, fissures, rectal exam if needed, frequency of stooling, quality of stool, rectal bleeding, other possible associated symptoms such as reflux/dyspepsia, vomiting, headaches, increase or decrease in appetite; 3) behavioral techniques, such as toileting after meal times, and other strategies are added; and 4) medicine and dietary adjustments are made. At each visit, the following instruments/questionnaires will be administered by a clinical psychologist: 1) social responsiveness scale; 2) Kaufman Brief Intelligence Test; 3) Child Behavior Checklist; 4) Aberrant Behavior Checklist; 5) Pediatric Quality of Life Inventory (Peds QL); 6) Repetitive Behavioral Scale-Revised; 7) Autism Impact Measure; 8) Pearson Short Sensory Profile. The Vineland will be administered at baseline and 12 months. The ADOS-2 will be used at baseline to ensure an ASD diagnosis.

At each visit, subject urine is collected and stored until an assay for the oxidative stress marker F2-isoprostane is measured.

A buccal swab is collected and DNA extracted for future genetic studies.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking of any ethnicity
* Boys or girls aged 5 years 0 months to 17 years 11 months

  * A clinical diagnosis of functional constipation (FC) for the ASD+/FC+ group, with or without encopresis
  * Clinical assessment of ASD using Diagnostic and Statistical Manual of Mental Disorders (DSM IV or V criteria)
  * ADOS-validated diagnosis of ASD
* Gestational age between 36 and 42 weeks
* Birth weight of at least 2500 grams

  * Children with suspected or an existing clinical diagnosis of ASD and FC will be recruited and consented for the study. Assessments and clinical diagnosis may be completed and confirmed through the Baseline study visit for subjects to be eligible.

    * Teacher participation is not required for child participation. However, teacher participation will be requested around the time of child enrollment.

Exclusion Criteria:

* Severe sensory or motor impairments (deafness, blindness;
* Identified inherited metabolic, syndromic, or progressive neurological disorders (including epilepsy, Down Syndrome, Rett Syndrome, Tuberous Sclerosis, Neurofibromatosis, Fragile X Syndrome);
* A non-functional GID, such as ulcerative colitis, Celiac disease or Hirschsprung's disease;
* Failure to meet birth weight/gestational age as noted above
* Participation in another ASD research study at the same time
* Not enrolled in an ASD intervention program

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Autism Spectrum Disorders with and without functional constipation
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Reduction in F2-IsoProstanes (IsoPs) oxidative stress biomarker | 1 year
Reduction in T-score from Social Responsiveness Scale (SRS-2) (Teacher questionnaire) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pat Levitt, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - The Center for Autism & Neurodevelopmental Disorders, Santa Ana, California

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT02442115/Prot_SAP_001.pdf